CLINICAL TRIAL: NCT02697344
Title: Phase I/II Trial of AT-101 in Combination With Lenalidomide and Dexamethasone in Patients With Relapsed Symptomatic Multiple Myeloma
Brief Title: Gossypol Acetic Acid With Lenalidomide and Dexamethasone in Treating Patients With Relapsed Symptomatic Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1384B; NCI-2016-00073 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 15-003501 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2016-02-22; First posted 2016-03-03 (Estimated); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Recurrent Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Lenalidomide; gossypol acetic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (AT-101, lenalidomide, and dexamethasone) (Experimental): Patients receive R-(-)-gossypol acetic acid PO QD on days 1-21. Beginning in course 2, patients also receive lenalidomide PO QD on days 1-21 and dexamethasone PO QD on days 1, 8, and 15 of courses 2-12. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dexamethasone; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide; Other: Pharmacological Study; Drug: R-(-)-Gossypol Acetic Acid

INTERVENTIONS:
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Other: Pharmacological Study — Correlative studies
Drug: R-(-)-Gossypol Acetic Acid — Given PO
  Other Names: (-)-Gossypol Acetic Acid; AT-101; GOSSYPOL ACETIC ACID, (R)-

SUMMARY:
This phase I trial studies the side effects and best dose of R-(-)-gossypol acetic acid when given together with lenalidomide and dexamethasone and to see how well it works in treating patients with multiple myeloma, also known as plasma cell myeloma, that has come back after a period of improvement or has gotten worse after treatment. R-(-)-gossypol acetic acid may stop the growth of cancer cells by recognizing certain proteins and stimulating programmed cell death. Lenalidomide may stimulate or suppress the immune system in different ways and stop cancer cells from growing. Drugs used in chemotherapy, such as dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving R-(-)-gossypol acetic acid with lenalidomide and dexamethasone may work better in treating patients with multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose of R-(-)-gossypol acetic acid (AT-101) that can be combined with lenalidomide and dexamethasone in patients with relapsed symptomatic multiple myeloma (MM). (Phase I) II. To determine the overall response rate (partial response or better) of AT-101 when used in combination with lenalidomide and dexamethasone in patients with relapsed symptomatic MM. (Phase II)

SECONDARY OBJECTIVES:

I. To determine the progression free survival and overall survival among patients with relapsed symptomatic MM following treatment with AT-101 in combination with lenalidomide and dexamethasone.

II. To determine the toxicities associated with AT-101 in combination with lenalidomide and dexamethasone in patients with relapsed symptomatic MM.

TERTIARY OBJECTIVES:

I. Determine in vivo the anti-myeloma effect of AT-101 alone by assessing extent of decrease in M-protein (serum and/or urine) after 1 cycle of AT-101 alone.

II. Determine the pharmacodynamics effect of AT-101 in combination with lenalidomide and dexamethasone treatment on primary myeloma cell in vivo.

III. Explore potential mechanism of resistance to AT-101 in combination with lenalidomide and dexamethasone therapy and the role of B-cell CLL/lymphoma 2 (Bcl-2).

OUTLINE: This is a phase I dose-escalation study of R-(-)-gossypol acetic acid followed by a phase II study.

Patients receive R-(-)-gossypol acetic acid orally (PO) once a day (QD) on days 1-21. Beginning in course 2, patients also receive lenalidomide PO QD on days 1-21 and dexamethasone PO QD on days 1, 8, and 15. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Calculated creatinine clearance (using Cockcroft-Gault equation) >= 60 mL/min =<14 days prior to registration
* Absolute neutrophil count (ANC) >= 1000/mm^3 =<14 days prior to registration
* Platelet count >= 75000/mm^3 =<14 days prior to registration
* Hemoglobin >= 8.0 g/dL =<14 days prior to registration
* Patient must have relapsed and symptomatic multiple myeloma
* Measurable disease of multiple myeloma as defined by at least ONE of the following:

  * Serum monoclonal protein >= 1.0 g/dL
  * >= 200 mg of monoclonal protein in the urine on 24 hour electrophoresis
  * Serum immunoglobulin free light chain >= 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Patients must have received ≥3 prior regimens for multiple myeloma
* Provide informed written consent
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Arm A Only (Closed): Willing to provide bone marrow and blood samples for correlative research purposes

Exclusion Criteria:

* Monoclonal gammopathy of undetermined significance (MGUS) or smoldering myeloma
* Patients who received daratumumab, pomalidomide and dexamethasone as the most immediate prior line of therapy prior to trial enrollment (prior therapy with a daratumumab-based or a pomalidomide-based regimen are allowed and prior daratumumab-pomalidomide-dexamethasone is allowed so long as it was not given as the most immediate prior line of therapy prior to trial enrollment).
* Other malignancy requiring active therapy EXCEPTIONS: non-melanotic skin cancer or carcinoma-in-situ of the cervix; NOTE: if there is a history of prior malignancy, they must not be receiving other specific treatment for their cancer
* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens (e.g., uncontrolled infection, uncompensated heart or lung disease)
* Other concurrent chemotherapy, radiotherapy, or any ancillary therapy considered investigational; NOTE: Bisphosphonates are considered to be supportive care rather than therapy, and are thus allowed while on protocol treatment
* Prior severe skin reaction (toxic epidermal necrosis) with immunomodulating agents
* Major surgery =< 14 days before study registration
* Concurrent medical problems that preclude use of deep vein thrombosis (DVT) prophylaxis with lenalidomide treatment
* Evidence of current uncontrolled cardiovascular conditions, including cardiac arrhythmias, congestive heart failure, angina, or myocardial infarction =< 6 months prior to registration
* Immunocompromised patients and patients known human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy NOTE: Patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial
* Uncontrolled intercurrent illness including, but not limited to

  * ongoing or active infection
  * symptomatic congestive heart failure
  * unstable angina pectoris
  * cardiac arrhythmia
  * or psychiatric illness/social situations that would limit compliance with study requirements
* Known allergy to any of the study medications, their analogues or excipients in the various formulations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-04-14 (Actual); Primary Completion 2018-10-26 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Maximally tolerated dose of AT-101 in combination with lenalidomide and dexamethasone defined as the dose level below the lowest dose that induces dose-limiting toxicity in at least one-third of patients (Phase I) | Up to day 28 of course 2
  The number and severity of all adverse events (overall and by dose-level) will be tabulated and summarized in this patient population. The Grade 3+ adverse events will also be described and summarized in a similar fashion.
Overall response rate, with response defined to be a stringent complete response, complete response, very good partial response, or partial response (Phase II) | Up to 3 years
  Responses will be summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease in this patient population. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 30 days after the last day of study drug treatment
  The maximum grade for each type of adverse event, regardless of causality, will be recorded and reported for each patient, and frequency tables will be reviewed to determine adverse event patterns.
Overall survival (Phase II) | Time from registration to death due to any cause, assessed up to 3 years
  Estimated using the method of Kaplan-Meier.
Progression free survival (Phase II) | Time from registration to the earliest date of documentation of disease progression or death due to any cause, assesse up to 3 years
  Estimated using the method of Kaplan-Meier.

OTHER OUTCOMES:
Biochemical response, measured by change in serum/urine M-proteins and light chains | Baseline to day 28 of course 1
  The degree of response of these tumor biomarkers will be evaluated (percentage and absolute decrease)
Change in basal expression of Bcl-2 and its family members | Baseline to after completion of 2 courses of treatment (56 days)
  Basal expression will be summarized descriptively for each target. Changes in expression over time will be evaluated for each target using Wilcoxon's signed rank test.
Change in basal expression pattern of protein kinase B (Akt), mitogen-activated protein kinase 1 (Erk), and mitogen-activated protein kinase (MAPK) | Baseline to after completion of 2 courses of treatment (56 days)
  Basal expression will be summarized descriptively for each target. Changes in expression over time will be evaluated for each target using Wilcoxon's signed rank test
Change in Cereblon expression | Baseline to time of relapse/resistance (relapse after a clinical response or progressive disease while on therapy, up to 3 years)
  Analyzed to determine if clinical response to lenalidomide/dexamethasone is linked to Cereblon expression. The expression will be summarized descriptively.
Resistance to AT-101, measured by change in basal Bcl-2 and Mcl-2 binding domain sequence | Baseline to time of relapse/resistance (up to 3 years)
  These targets will be summarized descriptively. The baseline values will be compared with the values at the time of relapse/resistance using Wilcoxon's signed rank test.
Resistance to lenalidomide/dexamethasone, measured by change in expression of signaling molecules Akt, Erk1/2, and MAPK | Baseline to time of relapse/resistance (up to 3 years)
  Comparison will be drawn between the pre-treatment samples and those obtained at time of resistance using Wilcoxon's signed rank test. Correlation will be made with clinical response to therapy (responder vs. non-responder) using Wilcoxon's rank sum test.

CONTACTS AND LOCATIONS:
Overall Officials: Sikander Ailawadhi, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials